CLINICAL TRIAL: NCT03460236
Title: Precision Assessment of Platelet Rich Plasma for Joint Preservation
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F2452-R; 43655 (Other: IRB protocol number)
Record Dates: First submitted 2018-01-10; First posted 2018-03-09 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis
Keywords: PRP; osteoarthritis; MRI; gait; patient reported outcome
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One tube of blood identified with a unique number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PRP: Symptomatic early knee osteoarthritis subjects who have elected to receive PRP treatment.

SUMMARY:
Knee Osteoarthritis (OA) is a leading cause of premature disability in Veterans who develop knee OA at higher rates and younger ages than the population in general. For those with symptomatic early knee OA, who are years to decades away from meeting clinical indications for knee replacement surgery, knee injections have been a key treatment option. In recent years, platelet rich plasma (PRP) injections have gained increasing attention for improving pain and function in patients with knee OA. Basic science studies also suggest that PRP may also potentially stimulate repair responses to articular cartilage. However, the mechanisms of action of PRP in the treatment of knee OA are unknown. Because autologous blood is used, the PRP composition differs between patients. It is also unknown whether these differences in PRP composition affect clinical outcomes. This study will address these gaps and provide critical new and objective information on PRP treatment effects in Veterans and additional women with early knee OA important to improving clinical use of this new treatment.

DETAILED DESCRIPTION:
Because very little is known about either the mechanisms of action or objective clinical outcomes of PRP treatment for knee OA, the investigators propose a prospective "pre-post" study that will permit us to identify areas where more rigorous clinical outcomes and mechanistic research may be warranted. The proposed work includes special elements of: (1) quantitative metrics to assess clinical outcomes, (2) correlation of candidate beneficial proteins with clinical outcomes, and (3) proteomic evaluation of the injected PRP. This work will use an innovative multi-disciplinary, personalized approach to evaluate the effects of PRP composition on both function, as assessed by patient-reported outcomes and gait analysis, and cartilage matrix structure as assessed by quantitative MRI

ELIGIBILITY:
Inclusion Criteria:

* symptomatic early knee OA
* full weight-bearing status
* have elected to receive PRP treatment
* Male veterans
* Female veterans

Exclusion Criteria:

* inflammatory arthritis, gout or recurrent pseudogout
* symptomatic OA of other lower extremity joints
* BMI >35 kg/m2
* use of walking, orthopedic, or prosthetic assistive device
* severe systemic disease defined as American Society of Anesthesiologists (ASA) 3 or above56
* inability to have MRI
* pregnant or intending to become pregnant during the study
* predominantly patellofemoral disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic early knee osteoarthritis subjects who have elected to receive PRP treatment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance R. Chu, MD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silva MDC, Perriman DM, Fearon AM, Couldrick JM, Scarvell JM. Minimal important change and difference for knee osteoarthritis outcome measurement tools after non-surgical interventions: a systematic review. BMJ Open. 2023 May 18;13(5):e063026. doi: 10.1136/bmjopen-2022-063026. PMID 37202126

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, 16 failed radiographic screening before assignment to the study.
Groups:
- Platelet Rich Plasma: Symptomatic early knee osteoarthritis subjects who have elected to receive PRP treatment.
Period: Overall Study
Arm/Group | Platelet Rich Plasma
Started | 90
Completed | 63
Not Completed | 27
Not completed — failed radiographic screening | 16
Not completed — Withdrawal by Subject | 11

BASELINE CHARACTERISTICS:
Population: Males and females with early knee osteoarthritis pain.
Groups:
- Platelet Rich Plasma Injection Group: Symptomatic early knee osteoarthritis subjects who have elected to receive PRP treatment.
Arm/Group | Platelet Rich Plasma Injection Group
Number analyzed (Participants) | 90
Age, Continuous [Mean (Full Range); unit: years] | 55 [30 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 68
  More than one race | 1
  Unknown or Not Reported | 5
Body Mass Index [Mean (Full Range); unit: kg/m²] | 27.78499 [20.92132184 to 35.2026893]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Knee Pain Improvement Over 6 Months Following PRP Injections
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain scores were determined through standardized questionnaires to evaluate osteoarthritis of the knee. The KOOS Pain scale consists of 9 questions with each response valued on an ordinal scale 0-4. KOOS Pain scores are transformed so that higher scores indicate less pain. Successful pain improvement is determined from the number of participants with changes in KOOS Pain in excess of the previously determined threshold of 12.4pts for minimal important change after non-surgical intervention for knee pain.
Time Frame: Baseline to 6 months
Population: The 63 participants who completed both baseline and 6-month follow-up patient reported outcome surveys.
Measure: Count of Participants; unit: Participants
Groups:
- Platelet Rich Plasma (PRP) Recipients: Symptomatic early knee osteoarthritis subjects who have elected to receive PRP treatment.
Arm/Group | Platelet Rich Plasma (PRP) Recipients
Number analyzed (Participants) | 63
Participants | 25

2. Primary Outcome: Number of Participants With Successful Knee Function Improvement Over 6 Months Following PRP Injections
Description: Knee Function was determined from Western Ontario and McMaster University Osteoarthritis Index (WOMAC) scores, standardized questionnaires to evaluate osteoarthritis of the knee. The WOMAC Function scale consists of 17 questions, with each response valued on an ordinal scale of 0-4. Higher numbers indicate more physical disability. Successful functional improvement is determined from the number of participants with changes in the WOMAC Function score in excess of the previously determined threshold of -17pts for minimal important functional change after non-surgical intervention.
Time Frame: Baseline to 6 months
Population: The 63 participants who completed both baseline and 6-month follow-up patient reported outcome surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet Rich Plasma (PRP) Recipients
Number analyzed (Participants) | 63
Participants | 12

ADVERSE EVENTS:
Time Frame: 6 months
Description: The principal investigator and team followed participants for 6 months and reported adverse events to the IRB immediately, if there were any.
Arm/Group | Platelet Rich Plasma (PRP) Recipients
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT03460236/Prot_SAP_ICF_000.pdf